CLINICAL TRIAL: NCT03607838
Title: A Multicenter, Randomized, Double-blind, Sham-controlled, Comparative Study of SI-6603 in Subjects With Lumbar Disc Herniation (Phase 3)
Brief Title: SI-6603 (Condoliase) Study for Lumbar Disc Herniation (Discovery 6603 Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6603 /1133
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar disc herniation; Radiculopathy; Sciatica; Intradiscal injection; Chemonucleolysis
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy; Sciatica | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SI-6603 (Experimental): Condoliase: 1.25U, intradiscal injection, one time
  For patients in the active treatment group, a volume of 1.0 mL was administered into the intervertebral disc in a single dose.
  Interventions: Drug: SI-6603
- Sham (Sham Comparator): Sham injection
  For patients in the control group, a solution was not prepared and the needle was not placed in the intervertebral disc.
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: SI-6603 — SI-6603 will be injected into an intervertebral disc.
  Arms: SI-6603
Drug: Sham injection — The injection will be performed without needle placement into an intervertebral disc.
  Arms: Sham

SUMMARY:
This study is to evaluate the effectiveness of a single-dose intervertebral disc injection of SI-6603 in subjects with lumbar disc herniation (LDH)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with single-level LDH (L4-L5 or L5-S1 (or L5-L6)) with clear, demonstrable nerve root impingement as assessed by magnetic resonance imaging (MRI) and clinical symptoms corresponding to position of the impaired nerve root.
* Subjects with radiculopathy/radicular leg pain in the unilateral leg for 6 weeks or more but 1 year or less.
* Subjects with positive result of Straight Leg Raise (SLR) test (≤70°) only on the ipsilateral leg having chief complaint of radiculopathy
* Subjects with inadequate improvement in pain caused by LDH despite 6 weeks or more of conservative treatment.

Exclusion Criteria:

* Subjects who have 2 or more lumbar disc herniations as assessed by MRI.
* Subjects who have undergone a lumbar operation, lumbar percutaneous nucleotomy, or lumbar intradiscal therapies at the affected level of lumbar spine.
* Subjects who have received block procedure (e.g., spinal injection, epidural injection or nerve block) for treatment of LDH, oral or injectable corticosteroids within 28 days prior to randomization.
* Subjects who have received opioids or cannabis by any route of administration, local anesthesia to the back, buttock, or posterior/lateral aspects of the affected leg within 7 days prior to randomization.
* Subjects with a body mass index (BMI) ≥40.
* Subjects who are receiving compensation according to the Workers' Compensation Act or are involved in personal injury litigation due to a lumbar-related injury.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (67):
  - Delta Clinical Research, Mobile, Alabama
  - Pain Medicine Associates, Inc., Fountain Valley, California
  - University of California San Diego - Center for Pain Medicine, La Jolla, California
  - The Helm Center for Pain Management, Laguna Woods, California
  - The Anand Spine Group, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Samaritan Center for Medical Research, Los Gatos, California
  - UC Davis Spine Center, Sacramento, California
  - Source Healthcare, Santa Monica, California
  - Boulder Neurosurgical Associates, Boulder, Colorado
  - DBPS Research, LLC, Greenwood Village, Colorado
  - International Spine, Pain, and Performance Center, Washington D.C., District of Columbia
  - Florida Spine Institute, Clearwater, Florida
  - Spine and Orthopedic Center, Deerfield Beach, Florida
  - Deland Clinical research Unit, DeLand, Florida
  - Science Connections, LLC, Doral, Florida
  - Coastal Clinical Research, Fernandina Beach, Florida
  - Holy Cross Medical Group, Fort Lauderdale, Florida
  - Coastal Clinical Research, Jacksonville, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - Science Connections, LLC (Kendall), Miami, Florida
  - AMPM Research Clinic, Miami Gardens, Florida
  - Pain Relief Centers, St. Petersburg, Florida
  - Pain Relief Centers, Sun City Center, Florida
  - Tampa Pain Relief Center, Tampa, Florida
  - Florida Pain Relief Group, PLLC, Tampa, Florida
  - Premier Medical Associates, The Villages, Florida
  - Conquest Research, Winter Park, Florida
  - Augusta University - Medical College of Georgia, Augusta, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Injury Care Research, Boise, Idaho
  - Millennium Pain Center, Bloomington, Illinois
  - Chicago Anesthesia Pain Specialists, Chicago, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Neuroscience Research Center LLC, Overland Park, Kansas
  - OtriMed Clinical Research, Edgewood, Kentucky
  - Clinical Trials of Southwest Louisiana, LLC, Lake Charles, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - St. Louis Pain Consultants, Chesterfield, Missouri
  - Comprehensive and Interventional Pain Management LLP, Henderson, Nevada
  - Innovative Pain Care Center, Las Vegas, Nevada
  - Interventional Spine Medicine, Barrington, New Hampshire
  - New Jersey Regenerative Institute, Cedar Knolls, New Jersey
  - New York - Presbyterian Queens, Flushing, New York
  - Drug Trials America, Hartsdale, New York
  - Ainsworth Institute Of Pain Management, New York, New York
  - University of Rochester- Neuromedicine Pain Management Center, Rochester, New York
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Clinical Inquest Center Ltd, Beavercreek, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - Medical Research International, Oklahoma City, Oklahoma
  - Oklahoma City Clinical Research Center, Oklahoma City, Oklahoma
  - Main Line Spine, King of Prussia, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - SC Pain & Spine Specialists, Murrells Inlet, South Carolina
  - Ascension Spine and Scoliosis Center, Austin, Texas
  - HRMD Research, Dallas, Texas
  - Advanced Medical Trials, Georgetown, Texas
  - Interventional Pain Specialists, Pasadena, Texas
  - ARH Research, LLC., The Woodlands, Texas
  - JBR Clinical Research, Salt Lake City, Utah
  - University of Virginia Orthopaedic Spine Center, Charlottesville, Virginia
  - Virginia iSpine Physicians, P.C., Richmond, Virginia
  - Gershon Pain Specialists, Virginia Beach, Virginia
  - Swedish Pain Management, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Derived] Macadaeg KE, Kim KD, Gupta PB, Rivera J, Patel A, Chauhan K, Watanabe J, Seo T, Zucker E, Candido K. Impact of Condoliase on Health-related Quality of Life in Participants With Radicular Leg Pain Associated With Lumbar Disk Herniation: Results From a United States Phase 3 Clinical Trial. Spine (Phila Pa 1976). 2025 Jun 15;50(12):796-803. doi: 10.1097/BRS.0000000000005327. Epub 2025 Mar 11. PMID 40066868
- [Derived] Kim KD, Ahadian F, Hassanzadeh H, Rivera J, Candido K, Gershon S, Patel A, Gupta PB, Miller AE, Formoso FJ, Fuerst T, Zucker E, Seo T, Watanabe J, Matsuyama Y, Chiba K, Macadaeg KE. A phase 3, randomized, double-blind, sham-controlled trial of SI-6603 (condoliase) in patients with radicular leg pain associated with lumbar disc herniation. Spine J. 2024 Dec;24(12):2285-2296. doi: 10.1016/j.spinee.2024.08.006. Epub 2024 Aug 19. PMID 39168360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty sites screened at least 1 subject, and 41 of these sites enrolled at least 1 subject. The first participant was enrolled in November 2018 and the last participant was enrolled in March 2022.
Pre-assignment Details: A total of 807 subjects were screened for enrollment. Of the 352 subjects randomized in the study, 176 were randomized to the SI-6603 group and 176 were randomized to the sham control group. Study drug was received by 169 SI-6603 subjects, and 172 subjects underwent sham control. The reasons for discontinuation from the study before injection were 'withdrawal of consent' (4), 'failure to meet randomization criteria' (3), 'other' (3) and 'physician decision' (1).
Groups:
- Sham: Sham injection
  For patients in the control group, a solution was not prepared, and the needle was not placed in the intervertebral disc.
Period: Overall Study
Arm/Group | SI-6603 | Sham
Started (Randomized) | 176 | 176
Injected | 169 | 172
Evaluated Week 13 | 156 | 155
Completed (Week 52) | 135 | 130
Not Completed | 41 | 46
Not completed — Lack of Efficacy | 14 | 20
Not completed — Withdrawal by Subject | 13 | 8
Not completed — Lost to Follow-up | 6 | 11
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Failure to meet randomization criteria | 1 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Due to work | 1 | 0
Not completed — Litigation | 0 | 1
Not completed — Temperature excursion for study drug | 0 | 1
Not completed — Change of mind | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | SI-6603 | Sham | Total
Number analyzed (Participants) | 169 | 172 | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9.36) | 45.9 (9.84) | 46.3 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 83 | 157
  Male | 95 | 89 | 184
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 43 | 90
  Not Hispanic or Latino | 122 | 129 | 251
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 9 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 14 | 32
  White | 137 | 142 | 279
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 6 | 5 | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter] | 29.0 (4.92) | 28.4 (4.86) | 28.7 (4.89)
Smoking History [Count of Participants; unit: Participants]
  Never smoked | 106 | 103 | 209
  Past smoker | 34 | 36 | 70
  Current smoker | 29 | 33 | 62
Occupation [Count of Participants; unit: Participants]
  Heavy labor | 39 | 49 | 88
  Light labor | 130 | 123 | 253
Days of Onset of Current Leg Pain [Mean (Standard Deviation); unit: days] | 161.9 (83.57) | 172.2 (79.65) | 167.1 (81.66)
Herniation Site [Count of Participants; unit: Participants] — L4-L5=The disc between the 4th and 5th lumbar vertebra; L5-S1=The disc between the 5th lumbar vertebra and 1st sacral vertebra
  Participants
    L4-L5 | 70 | 71 | 141
    L5-S1 | 99 | 101 | 200
Worst Leg Pain (VAS) [Mean (Standard Deviation); unit: mm] — The average of worst leg pain score during the past 24 hours over the previous 7 days, as assessed by 100 mm Visual Analog Scale (VAS). VAS is a pain assessment tool with 0 mm representing an absence of pain, and 100 mm representing the worst pain patients have ever experienced.
  mm | 71.99 (9.554) | 71.82 (9.751) | 71.91 (9.640)
Worst Back Pain (VAS) [Mean (Standard Deviation); unit: mm] — The average of worst back pain score during the past 24 hours over the previous 7 days, as assessed by 100 mm Visual Analog Scale (VAS). VAS is a pain assessment tool with 0 mm representing an absence of pain, and 100 mm representing the worst pain patients have ever experienced.
  mm | 53.73 (25.250) | 52.45 (25.261) | 53.08 (25.227)
ODI score [Mean (Standard Deviation); unit: percentage of disability] — The Oswestry Disability Index (ODI) questionnaire is designed to provide information as to how the patient's back (or leg) pain affects their ability to manage in everyday life. A higher score on the ODI indicates a more severe disability. The final index score is calculated as a percentage, with 0% indicating no disability and 100% indicating highest disability.
  percentage of disability | 48.2 (11.77) | 49.1 (11.85) | 48.7 (11.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 13 in Average Worst Leg Pain Score During the Past 24 Hours Over the Previous 7 Days
Description: The primary endpoint was the change from baseline to Week 13 in average worst leg pain score during the past 24 hours over the previous 7 days, as assessed by 100 mm Visual Analog Scale (VAS). VAS is a pain assessment tool with 0 mm representing an absence of pain, and 100 mm representing the worst pain patients have ever experienced.
Time Frame: baseline and 13 weeks
Population: Modified intention-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SI-6603 | Sham
Number analyzed (Participants) | 169 | 172
units on a scale | -41.7 (2.38) | -34.2 (2.36)
Statistical Analysis 1: Comparison: SI-6603 vs Sham; Test type: Superiority; p = 0.0263, Mixed Models Analysis; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-14.1 to -0.9], Standard Error of Mean 3.35

2. Secondary Outcome: Change From Baseline to Week 52 in Average Worst Leg Pain Score During the Past 24 Hours Over the Previous 7 Days
Description: One of the key secondary endpoints was the change from baseline to Week 52 in average worst leg pain score during the past 24 hours over the previous 7 days, as assessed by 100 mm Visual Analog Scale (VAS). VAS is a pain assessment tool with 0 mm representing an absence of pain, and 100 mm representing the worst pain patients have ever experienced.
Time Frame: baseline and 52 weeks
Population: Modified intention-to-treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SI-6603 | Sham
Number analyzed (Participants) | 169 | 172
units on a scale | -51.2 (2.40) | -44.7 (2.41)
Statistical Analysis 1: Comparison: SI-6603 vs Sham; Test type: Superiority; p = 0.0558, Mixed Models Analysis — To control family-wise error rate for multiple tests of the primary and key secondary endpoints, serial gatekeeping testing algorithm was used; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-13.2 to 0.2], Standard Error of Mean 3.40

3. Secondary Outcome: Change From Baseline to Week 13 in Herniation Volume
Description: One of the key secondary endpoints was change from baseline to Week 13 in herniation volume. Herniation volumes were assessed with MRI by a central imaging facility.
Time Frame: baseline and 13 weeks
Population: Modified intention-to-treat population
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | SI-6603 | Sham
Number analyzed (Participants) | 169 | 172
mm^3 | -103.8 (10.74) | -78.1 (10.79)
Statistical Analysis 1: Comparison: SI-6603 vs Sham; Test type: Superiority; p = 0.0920, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -25.8, 95% CI 2-sided [-55.7 to 4.2], Standard Error of Mean 15.24

4. Secondary Outcome: Change From Baseline to Week 13 in Oswestry Disability Index (ODI) Score
Description: One of the key secondary endpioints was change from baseline to Week 13 in Oswestry Disability Index (ODI) score. The ODI questionnaire is designed to provide information as to how the patient's back (or leg) pain affects their ability to manage in everyday life. A higher score on the ODI indicates a more severe disability. The final index score is calculated as a percentage, with 0% indicating no disability and 100% indicating highest disability.
Time Frame: baseline and 13 weeks
Population: Modified intention-to-treat population
Measure: Least Squares Mean (Standard Error); unit: percentage of disability
Arm/Group | SI-6603 | Sham
Number analyzed (Participants) | 169 | 172
percentage of disability | -29.6 (1.38) | -25.4 (1.38)
Statistical Analysis 1: Comparison: SI-6603 vs Sham; Test type: Superiority; p = 0.0336, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-8.0 to -0.3], Standard Error of Mean 1.95

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The safety population was defined as all randomized subjects who received the study injection, analyzed according to the treatments subjects received. Two subjects who were randomized to SI-6603, received the sham. These two subjects were analyzed as part of the sham group for safety analyses.
Arm/Group | SI-6603 | Sham
All-Cause Mortality (participants affected / at risk) | 1/167 | 0/174
Serious Adverse Events (participants affected / at risk) | 7/167 | 6/174
Other Adverse Events (participants affected / at risk) | 91/167 | 62/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SI-6603 (N=167) | Sham (N=174)
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SI-6603 (N=167) | Sham (N=174)
Magnetic resonance imaging spinal abnormal (Investigations) | 47 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 13
Spinal X-ray abnormal (Investigations) | 13 | 3
COVID-19 (Infections and infestations) | 11 | 17
C-reactive protein increased (Investigations) | 10 | 6
Sciatica (Musculoskeletal and connective tissue disorders) | 6 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI do not make any publication of trial results without the written permission of sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT03607838/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT03607838/SAP_001.pdf